CLINICAL TRIAL: NCT01388023
Title: Phase 2 Clinical Study of a Day Long Effect of SmellX Palatal Patch Containing A Herbal Formula on Malodor
Brief Title: Day Long Prevention of Oral Malodor With a Palatal Patch (SmellX) Containing A Herbal Formula
Acronym: SmellX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Hadas Lamberg Dr., Hadassah Medical Centers
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1910552HMO-CTIL
Record Dates: First submitted 2008-01-17; First posted 2011-07-06 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Halitosis; Gingivitis
Keywords: SmellX; malodor; halitosis; herbal formulation; natural medicinals; slow release delivery system; gingivitis; Bad Breath
MeSH Terms: conditions — Halitosis; Gingivitis | interventions — Chlorhexidine; Listerine; diclosan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- smellx (Active Comparator): test group- SmellX palatal patch with the herbal formula
  Interventions: Dietary Supplement: herbal formula for fresh breath
- smellx palatal patch (Placebo Comparator): negative control group- SmellX palatal patch with out the herbal formula
  Interventions: Dietary Supplement: herbal formula for fresh breath
- chlorhexidine (Active Comparator): poositive control group-mouth wash with chlorhexidine 0.125%
  Interventions: Dietary Supplement: herbal formula for fresh breath
- listerine (Active Comparator): listerine mouth wash
  Interventions: Dietary Supplement: herbal formula for fresh breath

INTERVENTIONS:
Dietary Supplement: herbal formula for fresh breath — composition of herbal ingridients in a palatal mucoadhesive patch to remove volatile solfur compounds and reducequantity of vsc creating bacteria
  Other Names: chlorhexidine; listerine; diclosan

SUMMARY:
In a previous study the prevention of halitosis by the herbal formula and delivery system (SmellX), were established both in vitro and clinicaly. The duration of relief was established as long as 8 hours. In this study the investigators intend examine the day long efficacy of SmellX.

DETAILED DESCRIPTION:
Oral malodor is a common complaint among dental patients. This condition derives in most cases form the putrefactive activities of oral microorganisms, primarily anaerobic Gram negative bacteria. These bacteria reside on various locations within the oral cavity (e.g. tongue dorsum, interdental space, periodontal pockets, faulty and leaky restorations and tonsils) and breakdown salivary and oral proteins into their amino acid building blocks. Some of these amino acids (e.g. methionine and cysteine) are further metabolized yielding malodorous volatile sulfide compounds (VSC) such as methylmercaptan and hydrogen sulfide.The tongue dorsum and especially its posterior portion are considered the key location for this process. Therefore, the treatment regiment includes in most cases a daily use of tongue scrapers and mouthwashes. Indeed, a recent Cochrane systematic review found tongue scrapers to have short-term efficacy in controlling halitosis.

However, the use of tongue scrapers is unpleasant and induces in many cases a strong gag reflex, and apparently has very little effect on bacterial load of the tongue.

Furthermore, some mouthwashes have been shown to cause adverse side effects such as tooth staining. In a previous study we performed a set of related experiments on a new sustained release delivery system in the form of an adhesive tablet containing an herbal formulation. The adhesive tablet is applied to the palate. This places it right above, and in direct contact with the tongue dorsum, thus allowing a sustained release of the active ingredients directly to the target site. The ingredients of the herbal formulation have been previously shown to reduce malodor production in a salivary incubation assay. We tested the effect of this system on oral malodor production and VSC levels in a young healthy population, and the antimicrobial effect of its active ingredients on three known oral pathogens (Streptoccocus mutans, Porphyromonas gingivalis and Candida albicans. In this study we intend to examine a day long protocol to achieve a relief from oral halitosis for 24 houres.

ELIGIBILITY:
Inclusion Criteria:

* random gender
* age
* healthy people

Exclusion Criteria:

* used antibiotics in the last three months
* suffer from systemic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
reduction of VSC measurements with halimeter | 24 hr
  volatile solfur compounds can be measured with a halimeter as an indication of halitosis. decrease of vsc value from base line indicates success in reducing halitosis

SECONDARY OUTCOMES:
reduction of halitosis as measured by judge score | 24 hr
  judge score of halitosis on a scale of 1-5 is the gold standart for halitosis measurments. levels lower than base line indicate success in the treatment of halitosis

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Perez Davidi, DMD, Principal Investigator — Hadassah Medical Centers The hebrew university Jerusalem
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Background] Perez Davidi M, Beyth N, Sterer N, Feuerstein O, Weiss EI. Effect of liquid-polish coating on in vivo biofilm accumulation on provisional restorations: part 1. Quintessence Int. 2007 Jul-Aug;38(7):591-6. PMID 17694216
- [Result] Mizrahi B, Golenser J, Wolnerman JS, Domb AJ. Adhesive tablet effective for treating canker sores in humans. J Pharm Sci. 2004 Dec;93(12):2927-35. doi: 10.1002/jps.20193. PMID 15459950
- [Result] Sterer N, Rubinstein Y. Effect of various natural medicinals on salivary protein putrefaction and malodor production. Quintessence Int. 2006 Sep;37(8):653-8. PMID 16922026
- [Result] Sterer N. Antimicrobial effect of mastic gum methanolic extract against Porphyromonas gingivalis. J Med Food. 2006 Summer;9(2):290-2. doi: 10.1089/jmf.2006.9.290. PMID 16822220
- See also: Dr.Michael Perez Davidi — http://www.mypd.co.il